CLINICAL TRIAL: NCT05338450
Title: Clemastine Fumarate as Remyelinating Treatment in Internuclear Ophthalmoparesis and Multiple Sclerosis
Acronym: RESTORE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Sam Hof, MD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL78363.029.21; 2021-003677-66 (EudraCT Number)
Record Dates: First submitted 2022-04-06; First posted 2022-04-21 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis; Internuclear Ophthalmoplegia
Keywords: clemastine; fampridine; remyelination; eye-tracking; infrared oculography
MeSH Terms: conditions — Multiple Sclerosis; Ocular Motility Disorders | interventions — Clemastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clemastine Fumarate (Experimental)
  Interventions: Drug: Clemastine Fumarate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clemastine Fumarate — 4 mg of Clemastine Fumarate twice daily (8mg/day) orally for 6 months (180 days)
  Other Names: clemastine; Tavegyl
  Arms: Clemastine Fumarate
Drug: Placebo — Placebo equivalent to experimental arm
  Arms: Placebo

SUMMARY:
Rationale: Clemastine fumarate has been identified as potential remyelinating therapy for multiple sclerosis (MS). The (long-term) effects of clemastine need to be confirmed in clinical models for MS. Internuclear ophthalmoparesis (INO) may be used as a clinical model for investigating remyelinating therapies by measuring horizontal eye movements with infrared oculography. Furthermore, infrared oculography combined with a single dose of fampridine may be used to identify individuals with MS that are most likely to benefit from remyelinating therapy.

Objective: To assess the (long-term) efficacy of clemastine fumarate in improving dysconjugacy of eye movements in patients with internuclear ophthalmoparesis and multiple sclerosis. Secondly, to assess whether a response to a single dose of fampridine can predict the effects of clemastine treatment.

Study design: A single-centre double-blind randomized placebo-controlled trial consisting of a 6 months (180 days) treatment period followed by a 30 months follow-up period.

Study population: 80 MS patients, age 18-70 years, with INO.

Intervention: The intervention group will receive 4 mg of clemastine fumarate twice daily (8 mg/day) for 6 months (180 days), the control group will receive an equivalent amount of placebo. At baseline all participants will receive a single 10 mg dose of fampridine.

Main study parameters/endpoints: The primary outcome measure is the change in versional dysconjugacy index (VDI) of area under the curve (AUC) measured by infrared oculography. Secondary outcome measures include changes in other VDI measures (peak velocity per amplitude (PV/Am) and peak velocity (PV)), changes in VDI after single fampridine dose, other oculography parameters (e.g. saccadic latency, anti-saccades), (peripheral) retinal nerve fibre layer (pRNFL) and (macular) ganglion cell inner plexiform layer (mGCIPL) thickness measured by OCT, SDMT, EDSS, high and low contrast visual acuity, subjective visual functioning (NEI-VFQ-25 and NOV-AU questionnaire), quality of life (EQ5D-5L) and fatigue (CIS20R and NFI-MS questionnaire).

Nature and extent of the burden and risks: Participation in the study will consist of a total of 7 study visits. Study visits will include physical/neurological examination, infrared oculography, OCT, visual acuity tests, a cognition test (SDMT), 5 questionnaires and blood samples for safety laboratory tests. Considering both clemastine and fampridine are registered and well-established drugs and have been used in clinical practice, the estimated risk of unexpected adverse reactions is low.

ELIGIBILITY:
Inclusion criteria:

* A clinically definite diagnosis of multiple sclerosis.
* Diagnosis of internuclear ophthalmoparesis determined by the first infrared oculography at screening with either cut-off of 1.174 of the versional dysconjugacy index area under the curve (VDI-AUC) of 15° saccades or 1.180 of the versional dysconjugacy index peak velocity/saccadic amplitude (VDI-PV/Am) of 15° saccades.
* Age 18-70 (inclusive)
* Use of disease modifying therapies is not a contraindication.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent.

Exclusion criteria:

MS-related exclusion criteria:

* Changes in immunomodulatory therapy for multiple sclerosis in the 6 months before inclusion into the study.
* Clinical relapse of MS or high dosage corticosteroid use within 30 days before inclusion into the study.

IMP and medication related exclusion criteria:

* Contraindications to clemastine use, such as known porphyria or hypersensitivity to clemastine, other antihistamines with a similar chemical structure or any of the excipients.
* Contraindications to fampridine use, such as hypersensitivity to fampridine or any of the excipients, history of epilepsy, kidney disease (GFR <50 ml/min absolute contraindication; GFR = 50-80 ml/min relative contraindication), use of Organic Cation Transporter 2 (OCT2) inhibitors or history of significant cardiac arrhythmias or conduction block.
* Concomitant use of Fampridine or any other formulation of 4-aminopyridine (4AP) or diamino4ap that cannot be temporarily suspended prior to each study visit.
* Changes in the use of medication currently being investigated in remyelination trials within 6 months before screening, including but not limited to domperidone, liothyronine, quetiapine, testosterone and bazedoxifene.
* Non-incidental use of central nervous system depressants including but not limited to hypnotics, anxiolytics, monoamine-oxidase inhibitors (MAOI'S), tricyclic antidepressants, opioid analgesics and other antihistamines with sedating properties (e.g. promethazine).

Other medical history and concomitant disease exclusion criteria:

* History of significant cardiac conduction block.
* History of malignancy of any organ system (other than localized squamous or basal cell carcinoma of the skin or adequately treated cervical cancer), treated or untreated, within the past 3 years, regardless of whether there is evidence of local recurrence or metastases.
* Estimated glomerular filtration rate (eGFR) < 50 ml/min/1.73 m2; AST, ALT, or alkaline phosphatase > 2 times the upper limit of normal.
* Any ophthalmological disease which may prevent accurate infrared oculography assessment.
* Suicidal ideation or behaviour in 6 months prior to baseline.
* History of drug or alcohol abuse within the past year.
* Clinically significant cardiac, metabolic, hematologic, hepatic, immunologic, urologic, endocrinologic, neurologic, pulmonary, psychiatric, dermatologic, allergic, renal or other major diseases that in the PI's judgement may affect interpretation of study results or patient safety.
* History of or presence of clinically significant medical illness or laboratory abnormality that, in the opinion of the investigator would preclude participation in the study.

General exclusion criteria:

* Pregnancy at the time of inclusion into the study or planning on breastfeeding within the first 7 months after inclusion in the study.
* Involvement in other study protocol simultaneously without prior approval.
* Insufficient proficiency in reading Dutch.
* Unable or unwilling to suspend driving for a duration of 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Versional Dysconjugacy Index (VDI) - Area Under the Curve (VDI-AUC) (6 months) | 6 months
  Our main study parameter is the versional dysconjugacy index (VDI) measured by infrared oculography. The relative change in VDI from baseline will be compared between the treatment and control group at the end of treatment (6 months). The VDI of Area Under the Curve (AUC) will be our primary study parameter. This describes the area under the saccadic trajectory of the horizontal eye position.
Versional Dysconjugacy Index (VDI) - Area Under the Curve (VDI-AUC) (36 months) | 36 months
  The relative change in VDI from baseline will be compared between the treatment and control group at the end of follow-up (36 months).

SECONDARY OUTCOMES:
Other Versional Dysconjugacy Index (VDI) measures - Peak Velocity (VDI-pV + VDI-pV/Am) | 6 and 36 months
  Changes in other VDI measures (peak velocity (PV) and peak velocity divided by amplitude (PV/Am)).
Versional Dysconjugacy Index (VDI) - Response to Fampridine | Baseline
  Changes in VDI in response to single dose of Fampridine.
Other infrared oculography parameters - Saccadic Latency | 6 months and 36 months
  Changes in saccadic latency measured by infrared oculography.
Other infrared oculography parameters - Proportion of errors in an anti-saccadic task | 6 months and 36 months
  Changes in proportion of errors in an anti-saccadic task measured by infrared oculography.
Other infrared oculography parameters - Proportion of correct double-step saccades | 6 months and 36 months
  Changes in the proportion of correct double-step saccades measured by infrared oculography.
Other infrared oculography parameters - Error of the final eye position in double-step saccades | 6 months and 36 months
  Changes in the error of the final eye position in double-step saccades measured by infrared oculography.
Symbol Digit Modalities Test (SDMT) | 6 months and 36 months
Expanded Disability Status Scale (EDSS) | 6 months and 36 months
  Changes in the Expanded Disability Status Scale (EDSS), which ranges from 0 (normal neurological exam, no disability) to 10.0 (death due to MS).
High and Low Contrast Visual Acuity (HCVA and LCVA) | 6 months and 36 months
Subjective visual functioning (NEI-VFQ-25) | 6 months and 36 months
  Changes in subjective visual functioning measured by the National Eye Institute Visual Functioning Questionnaire - 25 (NEI-VFQ-25) questionnaire.
Visual complaints (NOV-AU) | 6 months and 36 months
  Changes in visual complaints measured by the Neuro-Ophthalmology Questionnaire Amsterdam UMC (NOV-AU) questionnaire.
Quality of life (EQ5D-5L) | 6 months and 36 months
  Changes in quality of life measured by EuroQol 5-Dimension 5-Level (EQ5D-5L) questionnaire.
Fatigue - CIS20R | 6 months and 36 months
  Prevalence and changes in fatigue measured by the Checklist Individual Strength (CIS20R) questionnaire.
Fatigue - NFI-MS | 6 months and 36 months
  Prevalence and changes in fatigue measured by the Neurological Fatigue Index MS (NFI-MS) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Petzold, Dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Hof S, van Rijn LJ, Uitdehaag BMJ, Nij Bijvank JA, Petzold A. Measuring and predicting the effect of remyelinating therapy in multiple sclerosis: a randomised controlled trial protocol (RESTORE). BMJ Open. 2024 Jan 30;14(1):e076651. doi: 10.1136/bmjopen-2023-076651. PMID 38296293